CLINICAL TRIAL: NCT01544114
Title: A 6-month, Multicenter, Open-label, Safety Study of VIMOVO (250 mg/20 mg, 375 mg/20 mg, and 500 mg/20 mg Naproxen/Esomeprazole) in Adolescents Aged 12 to 16 Years, Inclusive, With Juvenile Idiopathic Arthritis (JIA)
Brief Title: A Safety Study of VIMOVO in Adolescents With Juvenile Idiopathic Arthritis (JIA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1120C00037
Record Dates: First submitted 2012-02-21; First posted 2012-03-05 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Juvenile Idiopathic Arthritis (JIA)
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Naproxen; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VIMOVO (Experimental): Three VIMOVO strengths will be used in this study: 250 mg naproxen/20 mg esomeprazole magnesium (VIMOVO 250/20), 375 mg naproxen/20 mg esomeprazole magnesium (VIMOVO 375/20), and 500 mg naproxen/20 mg esomeprazole magnesium (VIMOVO 500/20). The VIMOVO strength allocated to each participant will be determined by the participant's weight at baseline and based on investigator's discretion.
  The target dose of the naproxen component will be within the range of 10-20 mg/kg/day divided twice daily (BID) with a maximum daily dose of 1000 mg.
  Interventions: Drug: VIMOVO 250/20; Drug: VIMOVO 375/20; Drug: VIMOVO 500/20

INTERVENTIONS:
Drug: VIMOVO 250/20 — 250 mg naproxen/20 mg esomeprazole magnesium oral tablet administered twice daily for up to 6 months
  Other Names: naproxen/esomeprazole
Drug: VIMOVO 375/20 — 375 mg naproxen/20 mg esomeprazole magnesium oral tablet administered twice daily for up to 6 months
  Other Names: naproxen/esomeprazole
Drug: VIMOVO 500/20 — 500 mg naproxen/20 mg esomeprazole magnesium oral tablet administered twice daily for up to 6 months
  Other Names: naproxen/esomeprazole

SUMMARY:
A 6-month study of the safety of VIMOVO in adolescents aged 12 to 16 years with JIA.

DETAILED DESCRIPTION:
Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian is able to provide written informed consent and patient is able to provide written assent if appropriate.
* Male and female adolescents aged 12 to 16 years at the time of enrollment.
* Diagnosed with JIA, including all the International League of Associations for Rheumatology JIA subtypes: oligoarthritis, polyarthritis (both rheumatoid factor [RF]+ and RF-), psoriatic arthritis, enthesitis-related arthritis, undifferentiated arthritis, and systemic arthritis.
* Based upon investigator judgment, it is determined appropriate for the patient to undergo 6 months of continuous treatment with VIMOVO.
* Body weight > 31 kg (68.2 lbs) and within the 5th to 95th percentile of body mass index for age.

Exclusion Criteria:

* In systemic JIA patients, presence of systemic features (ie, fever, rheumatoid rash, serositis, lymphadenopathy, macrophage activation syndrome) within 6 months prior to start of study drug.
* Currently taking (ie, within 4 weeks prior to start of drug) naproxen > 20 mg/kg/day or > 1000 mg total daily dose.
* Hemoglobin ≤ 8.5 g/dL.
* Individuals who have cardiovascular or cerebrovascular disease, based on history or risk factors.
* Any significant hepatic, renal, pulmonary, ophthalmologic, neurologic, or any other medical conditions indicated by medical/surgical history, physical, or laboratory examination that might put the patient at greater risk during the study.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2012-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- United States (17):
  - Research Site, Little Rock, Arkansas
  - Research Site, San Francisco, California
  - Research Site, Aurora, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, West Palm Beach, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Omaha, Nebraska
  - Research Site, Brooklyn, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Fairfax, Virginia

REFERENCES:
- [Derived] Lovell DJ, Dare JA, Francis-Sedlak M, Ball J, LaMoreaux BD, Von Scheven E, Reinhardt A, Jerath R, Alpan O, Gupta R, Goldsmith D, Zeft A, Naddaf H, Gottlieb B, Jung L, Holt RJ. A 6-month, multicenter, open-label study of fixed dose naproxen/esomeprazole in adolescent patients with juvenile idiopathic arthritis. Pediatr Rheumatol Online J. 2018 Jun 26;16(1):41. doi: 10.1186/s12969-018-0260-y. PMID 29941047
- See also: Related Info — http://www.vimovo.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 51 participants signed informed consent; 5 participants were not assigned to treatment (eligibility criteria not fulfilled).
Groups:
- VIMOVO 250 mg/20 mg: 250 mg naproxen/20 mg esomeprazole magnesium oral tablet administered twice daily for up to 6 months
- VIMOVO 375 mg/20 mg: 375 mg naproxen/20 mg esomeprazole magnesium oral tablet administered twice daily for up to 6 months
- VIMOVO 500 mg/20 mg: 500 mg naproxen/20 mg esomeprazole magnesium oral tablet administered twice daily for up to 6 months
Period: Overall Study
Arm/Group | VIMOVO 250 mg/20 mg | VIMOVO 375 mg/20 mg | VIMOVO 500 mg/20 mg
Started | 4 | 20 | 22
Completed (completed study and received 6 months of study drug) | 3 (completed study and received 6 months of study drug) | 16 (completed study and received 6 months of study drug) | 17 (completed study and received 6 months of study drug)
Not Completed | 1 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Adverse Event | 1 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIMOVO 250 mg/20 mg | VIMOVO 375 mg/20 mg | VIMOVO 500 mg/20 mg | Total
Number analyzed (Participants) | 4 | 20 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (0.96) | 13.6 (1.47) | 13.8 (1.33) | 13.6 (1.37)
Age, Customized [Count of Participants; unit: Participants]
  Age Group: 12 years old | 2 | 7 | 4 | 13
  Age Group: 13 years old | 1 | 4 | 7 | 12
  Age Group: 14 years old | 1 | 2 | 2 | 5
  Age Group: 15 years old | 0 | 5 | 7 | 12
  Age Group: 16 years old | 0 | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 15 | 15 | 33
  Male | 1 | 5 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and TEAEs Leading to Discontinuation (DC) of Study Drug
Description: An AE is defined as the development of an undesirable medical condition or the deterioration of a preexisting medical condition, whether or not considered causally related to treatment. An SAE is defined as an AE occurring during any study phase (ie, run-in, treatment, washout, follow-up), that fulfils one or more of the following criteria: results in death; is immediately life-threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity; is a congenital abnormality or birth defect; is an important medical event that may jeopardize the participant or may require medical intervention to prevent one of the outcomes listed above. AEs were considered treatment-emergent if they occurred after the first dose of study drug. Events were categorized as mild, moderate, and severe; participants were represented only with the maximum reported intensity.
Time Frame: SAEs were collected from signing of informed consent through Month 6 (or end of treatment) plus 14 days. AEs were collected from administration of VIMOVO through Month 6 (or end of treatment) plus 14 days.
Population: Safety analysis set: all participants who received at least 1 dose of study drug; participants were categorized according to the treatment medication they actually took.
Measure: Number; unit: participants
Groups:
- Total: 250 mg naproxen/20 mg esomeprazole magnesium, 375 mg naproxen/20 mg esomeprazole magnesium, or 500 mg naproxen/20 mg esomeprazole magnesium oral tablet administered twice daily for up to 6 months
Arm/Group | VIMOVO 250 mg/20 mg | VIMOVO 375 mg/20 mg | VIMOVO 500 mg/20 mg | Total
Number analyzed (Participants) | 4 | 20 | 22 | 46
participants
  Any TEAE | 4 | 16 | 17 | 37
  Mild TEAE | 1 | 9 | 8 | 18
  Moderate TEAE | 3 | 6 | 9 | 18
  Severe TEAE | 0 | 1 | 0 | 1
  Any related TEAE | 1 | 6 | 4 | 11
  Any SAE | 0 | 1 | 0 | 1
  Any related SAE | 0 | 1 | 0 | 1
  Any TEAE leading to death | 0 | 0 | 0 | 0
  Any TEAE leading to DC of study drug | 1 | 1 | 2 | 4
  Any related TEAE leading to DC of study drug | 1 | 1 | 1 | 3

2. Secondary Outcome: Pharmacokinetics (PK) of Esomeprazole: Area Under the Concentration-Time Curve From the Time of Dosing to the Last Measurable Concentration (AUC[0-t])
Time Frame: pre-dose, and up to 3 hours post-dose
Population: PK Analysis Set: all participants who received at least 1 dose of study drug and had at least 1 post-baseline PK blood sample result and no protocol deviations that would have an impact on any PK assessment; participants were categorized according to the treatment medication they actually took.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*µmol/L
Arm/Group | VIMOVO 250 mg/20 mg | VIMOVO 375 mg/20 mg | VIMOVO 500 mg/20 mg | Total
Number analyzed (Participants) | 4 | 16 | 20 | 40
hr*µmol/L | 2.2 (92) | 1.3 (170) | 1.2 (150) | 1.3 (150)

3. Secondary Outcome: PK of Esomeprazole: Oral Plasma Clearance (CL/F)
Time Frame: pre-dose, and up to 3 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | VIMOVO 250 mg/20 mg | VIMOVO 375 mg/20 mg | VIMOVO 500 mg/20 mg | Total
Number analyzed (Participants) | 4 | 16 | 20 | 40
L/h | 27 (92) | 44 (170) | 47 (150) | 43 (150)

4. Secondary Outcome: PK of Esomeprazole: Absorption Rate Constant (Ka)
Time Frame: pre-dose, and up to 3 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h^-1
Arm/Group | VIMOVO 250 mg/20 mg | VIMOVO 375 mg/20 mg | VIMOVO 500 mg/20 mg | Total
Number analyzed (Participants) | 4 | 16 | 20 | 40
h^-1 | 2.8 (140) | 2.6 (83) | 4.1 (70) | 3.3 (84)

5. Secondary Outcome: PK of Esomeprazole: Oral Volume of Distribution (V/F)
Time Frame: pre-dose, and up to 3 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | VIMOVO 250 mg/20 mg | VIMOVO 375 mg/20 mg | VIMOVO 500 mg/20 mg | Total
Number analyzed (Participants) | 4 | 16 | 20 | 40
L | 28 (240) | 61 (120) | 57 (130) | 55 (130)

6. Secondary Outcome: PK of Naproxen: Trough Plasma Concentrations
Description: Trough concentration was defined as lowest plasma concentration from pre-dose to 3 hours post-dose, for each individual participant.
Time Frame: Month 1 and Month 3: pre-dose, and up to 3 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | VIMOVO 250 mg/20 mg | VIMOVO 375 mg/20 mg | VIMOVO 500 mg/20 mg
Number analyzed (Participants) | 4 | 17 | 20
µg/mL
  Month 1 | 63.09 (40.1) | 19.29 (1334.9) | 40.71 (277.3)
  Month 3: number analyzed (Participants) | 2 | 14 | 13
  Month 3 | 63.16 (67.3) | 33.91 (476.0) | 40.69 (325.4)

ADVERSE EVENTS:
Time Frame: SAEs were collected from signing of informed consent through Month 6 (or end of treatment) plus 14 days. AEs were collected from administration of VIMOVO through Month 6 (or end of treatment) plus 14 days.
Arm/Group | VIMOVO 250 mg/20 mg | VIMOVO 375 mg/20 mg | VIMOVO 500 mg/20 mg | Total
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/20 | 0/22 | 1/46
Other Adverse Events (participants affected / at risk) | 4/4 | 16/20 | 17/22 | 37/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIMOVO 250 mg/20 mg (N=4) | VIMOVO 375 mg/20 mg (N=20) | VIMOVO 500 mg/20 mg (N=22) | Total (N=46)
Hepatitis Acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIMOVO 250 mg/20 mg (N=4) | VIMOVO 375 mg/20 mg (N=20) | VIMOVO 500 mg/20 mg (N=22) | Total (N=46)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 3 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 4
Nausea (Gastrointestinal disorders) | 0 | 3 | 1 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 6 | 9
Sinusitis (Infections and infestations) | 0 | 1 | 4 | 5
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 3
Headache (Nervous system disorders) | 1 | 1 | 2 | 4
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 2 | 2
Tooth Infection (Infections and infestations) | 0 | 1 | 1 | 2
Bacterial Vaginosis (Infections and infestations) | 0 | 0 | 1 | 1
Fungal Infection (Infections and infestations) | 0 | 1 | 0 | 1
Helicobacter Infection (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 1
Localized Infection (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Otitis Media (Infections and infestations) | 0 | 0 | 1 | 1
Trichomoniasis (Infections and infestations) | 1 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Juvenile Idiopathic Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Tendon Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Eye Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Arachnoid Cyst (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Breast Mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Increased Tendency to Bruise (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Dry Eye (Eye disorders) | 0 | 0 | 1 | 1
Uveitis (Eye disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 2 | 2
Thirst (General disorders) | 0 | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1 | 2
Liver Function Test Abnormal (Investigations) | 0 | 1 | 0 | 1
Weight Decreased (Investigations) | 0 | 0 | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights .